CLINICAL TRIAL: NCT07057973
Title: The Effectiveness of Preoperative Iron Therapy in Improving Anemia After Multi-level Lumbar Fusion in the Elderly
Acronym: PITAMLFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xuanwu_DLD
Record Dates: First submitted 2025-06-02; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Ferric Carboxymaltose
MeSH Terms: interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Placebo treatment
- Ferric carboxymaltose (Experimental): Ferric carboxymaltose treatment
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — The experimental group was treated with 1000 mg of ferric carboxymaltose
  Arms: Ferric carboxymaltose

SUMMARY:
Preoperative iron therapy has important value in improving the outcomes after lumbar fusion surgery, but there is significant heterogeneity in both domestic and international studies. International studies provide high-level evidence-based evidence for intravenous iron, but lack spinal surgery-specific data; domestic studies focus on the comparison of iron types and the improvement of clinical practice, but high-quality evidence is still insufficient. At present, there are still few studies on preoperative iron therapy in the field of spinal surgery, especially its specific impact on the prognosis of patients after lumbar fusion surgery is still unclear. Therefore, it is particularly important to study the preoperative iron supplementation regimen for lumbar fusion surgery to improve the efficacy and safety. Through multidisciplinary collaboration and technological innovation, preoperative iron therapy is expected to become an important part of accelerated recovery after lumbar fusion surgery.

DETAILED DESCRIPTION:
Preoperative iron therapy has important value in improving the outcomes after lumbar fusion surgery, but there is significant heterogeneity in both domestic and international studies. International studies provide high-level evidence-based evidence for intravenous iron, but lack spinal surgery-specific data; domestic studies focus on the comparison of iron types and the improvement of clinical practice, but high-quality evidence is still insufficient. At present, there are still few studies on preoperative iron therapy in the field of spinal surgery, especially its specific impact on the prognosis of patients after lumbar fusion surgery is still unclear. Therefore, it is particularly important to study the preoperative iron supplementation regimen for lumbar fusion surgery to improve the efficacy and safety. Through multidisciplinary collaboration and technological innovation, preoperative iron therapy is expected to become an important part of accelerated recovery after lumbar fusion surgery.

This study aimed to investigate the correlation between ferric carboxymaltose and iron deficiency anemia (IDA) patients with or without concurrent iron therapy on hemoglobin changes, 90-day adverse events, and satisfactory health-related quality of life (HRQOL) indicators after multilevel lumbar spine fusion.

Outcome measures

1. Differences in hemoglobin and iron metabolism indicators (serum iron, ferritin, transferrin, transferrin saturation) levels on the 1st, 4th, 7th day after surgery and at discharge
2. Differences in the incidence of adverse events and length of hospital stay within 90 days after lumbar multilevel fusion surgery Any adverse event (AAE): serious or minor adverse event Serious adverse events (SAE): pulmonary embolism, wound infection, deep vein thrombosis, sepsis, myocardial infarction, neurological complications, delirium, septic shock, reoperation Minor adverse events (MAE): wound dehiscence, hematoma, other wound complications, acute kidney injury, blood transfusion, cerebrospinal fluid leak, urinary tract infection, pneumonia
3. Study-specific surveys conducted at the time of assessment included the following health status-related quality of life scores (HRQOL): Visual Analog Scale (VAS), Oswestry Disability Index (ODI), and EuroQol-5D (EQ-5D), 36-Item Short Form Health Survey (SF-36)

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent multi-segment lumbar spine surgery;
* IDA patients aged 65 years or older (male: Hb < 120g/dL; female: Hb < 110g/dL);
* All patients completed the relevant questionnaire survey;

Exclusion Criteria:

* Age less than 65 years old;
* Previous surgery for spinal tumors, trauma or infection;
* Inflammatory or immune diseases (such as rheumatoid arthritis or systemic lupus erythematosus), acute kidney injury, progressive cancer and porphyria cutanea tarda);
* Non-adjacent segment surgery;
* History of allergy to ferric carboxymaltose or any intravenous iron preparations, asthma, atopic dermatitis or allergy;
* Decompensated cirrhosis and microcytic anemia;
* Incomplete clinical data;

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
the levels of hemoglobin | on the first, fourth, and seventh days after surgery and at four weeks
  the levels of hemoglobin
the level of iron metabolism indicators (serum iron, ferritin, transferrin, and transferrin saturation) | on the first, fourth, and seventh days after surgery and at 4 weeks
  the level of iron metabolism indicators (serum iron, ferritin, transferrin, and transferrin saturation)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No